CLINICAL TRIAL: NCT02042300
Title: Evaluation of Effectiveness and Safety of XIENCE Xpedition/Alpine/Sierra in Routine Clinical Practice; A MULTICENTER, PROSPECTIVE OBSERVATIONAL STUDY
Brief Title: XIENCE Xpedition/Alpine/Sierra in Routine Clinical Practice
Acronym: IRIS XPEDITION
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2013-11
Record Dates: First submitted 2014-01-14; First posted 2014-01-22 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Percutaneous Transluminal Coronary Angioplasty; Coronary Artery Disease
Keywords: XIENCE Xpedition; Routine Clinical Practice; Alpine; Sierra
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IRIS-Xpedition/Alpine/Sierra Cohort: XIENCE Xpedition/Alpine/Sierra
  Interventions: Device: XIENCE Xpedition/Alpine/Sierra

INTERVENTIONS:
Device: XIENCE Xpedition/Alpine/Sierra

SUMMARY:
The purpose of this study is to evaluate effectiveness and safety of XIENCE Xpedition/Alpine/Sierra in Routine Clinical Practice

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Intervention with XIENCE Xpedition or Alpine or Sierra everolimus eluting coronary stent
* Agreed with written informed consent form

Exclusion Criteria:

* Intervention with XIENCE Xpedition or Alpine or Sierra everolimus eluting coronary stent and other drug eluting stent at the same time
* Life expectancy of 1year and under
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with XIENCE Xpedition or Alpine or Sierra stent
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Composite event rate | 1year
  Death, non fatal myocardial infarction, Target Vessel Revascularization

SECONDARY OUTCOMES:
All death | 5year
Cardiac death | 5year
Myocardial infarction | 5year
Composite event of death or myocardial infarction | 5year
Composite event of cardiac death or myocardial infarction | 5year
Target Vessel revascularization | 5year
Target lesion revascularization | 5year
Stent thrombosis by an Academic Research Consortium (ARC) criteria | 5year
Stroke | 5year
procedural success | 3day
  defined as less than 30% residual stenosis at the completion of procedure without death or Q wave myocardial infarction or urgent revascularization
  participants will be followed for the duration of hospital stay, an expected average of 3days.

CONTACTS AND LOCATIONS:
Locations (26):
- South Korea (26):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - ChonBuk National University Hospital, Jeonju
  - Kwangju Christian Hospital, Kwangju
  - Dong-A Medical Center, Pusan
  - Inje University HAEUNDAE Paik Hospital, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.